CLINICAL TRIAL: NCT07037693
Title: Prediction of Postoperative Outcomes After Rectal Resection by the Comprehensive Complication Index (CCI): A Retrospective Comparative Study
Brief Title: Prediction of Postoperative Outcomes After Rectal Resection by the Comprehensive Complication Index (CCI)
Status: Completed | Type: Observational
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Yanic Ammann, Principal Investigator, Cantonal Hospital of St. Gallen
Other Study IDs: CCI rectal resection
Record Dates: First submitted 2025-06-06; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Rectal Diseases
MeSH Terms: conditions — Rectal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCI
  Interventions: Diagnostic Test: Comprehensive complication index (CCI)
- CDC
  Interventions: Diagnostic Test: Clavien-Dindo-Classification (CDC)

INTERVENTIONS:
Diagnostic Test: Comprehensive complication index (CCI) — Comprehensive complication index (CCI)
  Groups: CCI
Diagnostic Test: Clavien-Dindo-Classification (CDC) — Clavien-Dindo-Classification (CDC)
  Groups: CDC

SUMMARY:
Postoperative complications after rectal resection can worsen the short-term postoperative outcomes and the long-term survival. This study aims to compare the comprehensive complication index (CCI) and the commonly used Clavien-Dindo classification (CDC) in predicting postoperative outcomes after rectal resection.

ELIGIBILITY:
Inclusion Criteria:

* All patients with rectal resection at the Cantonal Hospital of St.Gallen between 2012 and June 2024.

Exclusion Criteria:

* Missing CCI data
* Missing CDC data
* Incomplete 30-day follow-up
* Decline to have their information included in the scientific data analysis
* Age under 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with rectal resection at the Cantonal Hospital of St.Gallen between 2012 and June 2024.
Sampling Method: Non-Probability Sample
Enrollment: 958 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Periprocedural
  The predictive ability of the comprehensive-complication index and the Clavien-Dindo classification regarding the length of hospital stay after rectal resection will be compared through an area under the curve (AUC) analysis.

SECONDARY OUTCOMES:
30-day readmission rate | 30 days
  The predictive ability of the comprehensive-complication index and the Clavien-Dindo classification regarding the 30-day readmission rate after rectal resection will be compared through an area under the curve (AUC) analysis.
90-day mortality | 90 days
  The predictive ability of the comprehensive-complication index and the Clavien-Dindo classification regarding the 90-day mortality after rectal resection will be compared through an area under the curve (AUC) analysis.
Overall survival | 5 years
  The patients 5-year overall survival will be compared between patients with low comprehensive-complication index and high comprehensive-complication index. A high comprehensive-complication score was defined as a score above the median score of the patients with a Clavien-Dinco classification grad 3a complication.
Comprehensive measure | 30 days
  Evaluation of the comprehensive measure of the comprehensive-complications index through analysis of the number and severity of all complications for patients with multiple complications. Comparison of the range of the comprehensice complications-index score in patients with the same Clavien-Dindo classification.

CONTACTS AND LOCATIONS:
Locations (1):
- HOCH Health Ostschweiz, Kantonsspital St.Gallen, Sankt Gallen, St.Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No